CLINICAL TRIAL: NCT02220660
Title: A Single-blind, Randomised, Two-way Crossover Phase I Study to Assess Safety, Tolerability and Pharmacokinetics of the Fixed Dose Combination of BI 1744 CL Plus BI 54903 XX Via Respimat® B Versus the Free Combination of BI 1744 CL Via Respimat® A and BI 54903 XX Via Respimat® B in Healthy Male and Female Volunteers
Brief Title: Safety, Tolerability and Pharmacokinetics of the Fixed Dose Combination of BI 1744 CL Plus BI 54903 XX Via Respimat® B Versus the Free Combination of BI 1744 CL Via Respimat® A and BI 54903 XX Via Respimat® B in Healthy Male and Female Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 1256.2
Record Dates: First submitted 2014-08-19; First posted 2014-08-20 (Estimated); Last update posted 2014-08-20 (Estimated); Status verified 2014-08

CONDITIONS: Healthy
MeSH Terms: interventions — olodaterol

ARMS (2):
- Free dose combination (Active Comparator)
  Interventions: Drug: BI 1744 CL; Drug: BI 54903 XX
- Fixed dose combination (Experimental)
  Interventions: Drug: BI 1744 CL + BI 54903 XX FDC; Drug: Placebo

INTERVENTIONS:
Drug: BI 1744 CL
  Arms: Free dose combination
Drug: BI 54903 XX
  Arms: Free dose combination
Drug: BI 1744 CL + BI 54903 XX FDC
  Arms: Fixed dose combination
Drug: Placebo
  Arms: Fixed dose combination

SUMMARY:
The primary objective of this study was to compare the systemic exposure of BI 1744 BS and CD 1857 XX (the active metabolite of the pro-drug BI 54903 XX) at steady state following inhalation of the fixed dose combination (FDC) BI 1744 CL plus BI 54903 XX (as ethanolic solution for inhalation, EIS) with the systemic exposure following inhalation of the free dose combination of BI 1744 CL (as aqueous solution for inhalation, AIS) and BI 54903 XX (EIS), respectively, when administered once-daily via Respimat® Inhaler (Respimat® A for AIS and Respimat® B for EIS) for 14 days in healthy volunteers. Secondary objectives were: to compare exposure to BI 1744 BS and CD 1857 XX after a single dose of the BI 1744 CL/BI 54903 XX FDC and the free dose combination, respectively; to compare exposure to BI 54903 XX after a single dose and at steady state after multiple doses of the BI 1744 CL/BI 54903 XX fixed dose combination and the free dose combination, respectively; to compare the safety and tolerability of BI 1744 CL and BI 54903 XX when administered as BI 1744 CL/BI 54903 XX fixed dose combination and as the free dose combination, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females according to the following criteria: Based upon a complete medical history, including the physical examination, vital signs (Blood pressure (BP), Pulse rate (PR)), 12-lead Electrocardiogram (ECG), clinical laboratory tests
* Age >= 21 and <= 50 years
* BMI >= 18.5 and <= 29.9 kg/m2
* Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice (GCP) and the local legislation

Exclusion Criteria:

* Any finding of the medical examination (including BP, PR and ECG) deviating from normal and of clinical relevance
* Any evidence of a clinically relevant concomitant disease
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Surgery of the gastrointestinal tract (except appendectomy)
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of relevant orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of relevant allergy/hypersensitivity (including allergy to drug or its excipients)
* Intake of drugs with a long half-life (> 24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial
* Use of drugs which might reasonably influence the results of the trial based on the knowledge at the time of protocol preparation within 10 days prior to administration or during the trial
* Participation in another trial with an investigational drug within two months prior to administration or during the trial
* Smoker (> 10 cigarettes or > 3 cigars or > 3 pipes/day)
* Inability to refrain from smoking on trial days
* alcohol abuse (more than 40 g/day)
* Drug abuse
* Blood donation (> 100 mL within four weeks prior to administration or during the trial)
* Excessive physical activities (within one week prior to administration or during the trial)
* Any laboratory value outside the reference range that is of clinical relevance
* Inability to comply with dietary regimen of trial site

For female Subjects:

* Pregnancy
* Positive pregnancy test
* No adequate contraception (adequate contraception e.g. sterilization, intrauterine pessary (IUP), oral contraceptives)
* Inability to maintain this adequate contraception during the whole study period
* Lactation period

Exclusion criteria specific for this study due to the known class side effect profile of ß2-mimetics and inhaled corticosteroids:

* Asthma or history of pulmonary hyperreactivity
* Hyperthyreosis
* Allergic rhinitis in need of treatment
* Clinically relevant cardiac arrhythmia
* Bacterial and viral infections of the lung including tuberculosis

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2009-03; Primary Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
AUC0-t,ss (area under the concentration time curve of the analyte in plasma from 0 to time t at steady state) | up to 24 hours after drug administration
Cmax (maximum measured concentration of the analyte in plasma) | up to 24 hours after drug administration

SECONDARY OUTCOMES:
AUC0-t,ss (area under the concentration time curve of the analyte in plasma from 0 to time t at steady state) | up to 24 hours after drug administration
Cpre (pre-dose concentration of the analyte in plasma) | immediately before drug administration
AUCt1-t2 (area under the concentration time curve of the analyte in plasma over the time interval t1 to t2) | up to 24 hours after drug administration
AUC0-t (area under the concentration time curve of the analyte in plasma from 0 to time t) | up to 24 hours after drug administration
AUC0-tz (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the time of the last quantifiable data point) | up to 24 hours after drug administration
AUCτ (area under the plasma concentration-time curve over a uniform dosing interval τ) | up to 24 hours after drug administration
AUC0-∞ (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | up to 24 hours after drug administration
%AUCtz-∞(the percentage of the AUC0-∞that is obtained by extrapolation) | up to 24 hours after drug administration
tmax (time from dosing to the maximum concentration of the analyte in plasma) | up to 24 hours after drug administration
λz (terminal rate constant of the analyte in plasma) | up to 24 hours after drug administration
t½ (terminal half-life of the analyte in plasma) | up to 24 hours after drug administration
MRTih (mean residence time of the analyte in the body after inhaled administration) | up to 24 hours after drug administration
CL/F (apparent clearance of the analyte in the plasma after extravascular administration) | up to 24 hours after drug administration
Vz/F (apparent volume of distribution of the analyte during the terminal phase following an extravascular dose) | up to 24 hours after drug administration